CLINICAL TRIAL: NCT03425786
Title: Benign Paroxysmal Positional Vertigo (BPPV) Training for Sports Medicine Providers in a Pediatric Concussion Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Jacob Brodsky, Director of the Balance and Vestibular Program, Boston Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: IRB-P00025099
Record Dates: First submitted 2018-01-25; First posted 2018-02-08 (Actual); Last update posted 2024-11-25 (Actual); Status verified 2024-11

CONDITIONS: Benign Paroxysmal Positional Vertigo
MeSH Terms: conditions — Benign Paroxysmal Positional Vertigo

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early BPPV Management (Experimental): Diagnostic and treatment training for BPPV.
  Interventions: Behavioral: Diagnostic and treatment training
- Late BPPV Management (Active Comparator): Diagnostic training for BPPV. Sports Medicine providers will refer patients positive for BPPV to an Otolaryngologist at our institution for treatment.
  Interventions: Behavioral: Diagnostic training

INTERVENTIONS:
Behavioral: Diagnostic training — Training in the Dix-Hallpike maneuver and the supine head roll test to diagnose BPPV.
  Arms: Late BPPV Management
Behavioral: Diagnostic and treatment training — Training in the Dix-Hallpike maneuver and the supine head roll test to diagnose BPPV. Training in the Epley and Barbecue maneuvers to treat BPPV.
  Arms: Early BPPV Management

SUMMARY:
The investigators are training a group of four pediatric Sports Medicine providers in BPPV maneuvers. All four providers will be trained in the diagnostic maneuvers, and two will be randomly selected to also be trained in the treatment maneuvers. The providers will be encouraged to use the diagnostic maneuvers on all new concussion patients whose initial visit is within 28 days of their injury. They will complete a survey at the start and end of the study to determine if they thought the training affected their understanding of BPPV and confidence in managing it, as well as determine any challenges they faced with learning/administering the maneuvers. Additionally, the investigators will determine if the additional training impacts time to recovery from concussion, as well as determine potential risk factors for BPPV in concussion.

DETAILED DESCRIPTION:
Benign paroxysmal positional vertigo (BPPV) is a common disorder of the inner ear that causes episodes of vertigo. BPPV occurs as a result of displacement of otoliths from their position on the utricle into one of the semicircular canals. Posterior canal BPPV is diagnosed by performing the Dix-Hallpike maneuver, and lateral canal BPPV is diagnosed by performing the supine head roll test (Pagnini-McClure maneuver). Most cases of BPPV will resolve spontaneously, but this can take weeks to months without intervention, and approximately a third of cases will not resolve without treatment. Repositioning maneuvers, such as the Epley maneuver and Barbecue maneuver, move the otolith crystals out of the affected semicircular canal and back to their position on the utricle organ. Such maneuvers have been shown to be highly effective at resolving BPPV, and typically only 1-2 treatments are required.

BPPV most commonly occurs as an isolated spontaneous disorder, but it can also occur following a concussion. While the diagnosis and treatment of BPPV is a routine component of most Otolaryngology and Neurology training programs, it is not a component of most Sports Medicine training programs. It is also common that providers who are taught to diagnose BPPV do not know how to treat it. Furthermore, the role of BPPV in concussion recovery has not been well studied. Hoffer and colleagues found BPPV to be present in nearly a third of adult military patients with dizziness immediately following a concussion, and they found that these patients had rapid symptom resolution following repositioning maneuvers. The investigators recently found evidence of BPPV in 21% of patients referred to their pediatric vestibular program clinic for prolonged dizziness symptoms following a concussion. The majority of these patients were successfully treated with repositioning maneuvers following their first visit to the vestibular clinic, but that visit occurred at a mean of 4 months following their initial injury.

In order to determine if early recognition and management of BPPV will expedite recovery from concussion in affected patients, the investigators will train a group of four pediatric Sports Medicine providers in BPPV maneuvers. All four providers will be trained by Dr. Jacob Brodsky in the Dix-Hallpike and head roll maneuvers (BPPV diagnosis; Both Groups A & B), and two will be randomly selected to also be trained by Dr. Brodsky in the Epley and Barbecue maneuvers (BPPV treatment; Group A only). The providers will be encouraged to use the Dix-Hallpike and head roll maneuvers on all new concussion patients whose initial visit is within 28 days of their injury to determine if the patients have BPPV. Providers who have been trained in treatment maneuvers (Group A, Early BPPV Management) will be encouraged to perform them accordingly on any patients with positive diagnostic maneuvers. Providers who have not been trained in treatment maneuvers (Group B, Late BPPV Management) will refer patients with suspected BPPV to Dr. Brodsky for treatment, as is currently the routine. Patients are not being directly randomized and do not need to do anything beyond attend their regularly scheduled appointments.

The Sports Medicine providers will complete a source document after each visit to document which maneuvers were performed and if the patient has recovered from concussion. They will also complete a survey at the start and end of the study to determine if they thought the training affected their understanding of BPPV and confidence in managing it, as well as determine any challenges they faced with learning/administering the maneuvers. The patients managed by providers in Group A will then be compared to patients managed by providers in Group B by multiple variables, including their post concussion symptom scores (PCSS), time to clearance for return to play, and time to symptom resolution. The investigators will also compare patients who were diagnosed with BPPV to those who were not to evaluate for risk factors for post-concussion BPPV, including comparison of age, gender, migraine history, prior concussion history, and mode of injury.

ELIGIBILITY:
Inclusion Criteria:

• Sports Medicine providers at Boston Children's Hospital who see a high volume of concussion patients

Exclusion Criteria:

• None

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 221 (Actual)
Dates: Start 2021-09-29 (Actual); Primary Completion 2023-01-31 (Actual); Study Completion 2023-03-01 (Actual)

PRIMARY OUTCOMES:
Survey of level of confidence in managing BPPV in concussion patients | 1 year
  Providers will complete a survey before and after the study to assess if their level of confidence in managing BPPV in concussion patients has changed. Providers will rate their level of confidence from 1 to 10, with 1 meaning not at all confident and 10 meaning very confident.

SECONDARY OUTCOMES:
Time to recovery from concussion | 1 year
  A comparison of time to recovery from concussion in patients whose providers had diagnostic training versus patients whose providers had diagnostic and treatment training.
Mode of concussion | 1 year
  A comparison of concussion patients by mode of concussion to determine if mode of concussion is a potential risk factor for BPPV.
Site of impact | 1 year
  A comparison of concussion patients by site of impact to determine if site of impact is a potential risk factor for BPPV.
Sport played when concussion sustained | 1 year
  A comparison of concussion patients by which sport they were playing when the concussion was sustained to determine if certain sports are a potential risk factor for BPPV.
Number of lifetime concussions | 1 year
  A comparison of concussion patients by number of lifetime concussions to determine if number of lifetime concussions is a potential risk factor for BPPV.
History of migraine | 1 year
  A comparison of concussion patients by history of migraine to determine if history of migraine is a potential risk factor for BPPV.

CONTACTS AND LOCATIONS:
Overall Officials: Jacob R Brodsky, MD, Principal Investigator — Boston Children's Hospital
Locations (1):
- Boston Children's Hospital Waltham, Waltham, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Centers for Disease Control and Prevention (CDC). Sports-related recurrent brain injuries--United States. MMWR Morb Mortal Wkly Rep. 1997 Mar 14;46(10):224-7. PMID 9082176
- [Background] Meehan WP 3rd, Mannix RC, Stracciolini A, Elbin RJ, Collins MW. Symptom severity predicts prolonged recovery after sport-related concussion, but age and amnesia do not. J Pediatr. 2013 Sep;163(3):721-5. doi: 10.1016/j.jpeds.2013.03.012. Epub 2013 Apr 26. PMID 23628374
- [Background] Lau BC, Kontos AP, Collins MW, Mucha A, Lovell MR. Which on-field signs/symptoms predict protracted recovery from sport-related concussion among high school football players? Am J Sports Med. 2011 Nov;39(11):2311-8. doi: 10.1177/0363546511410655. Epub 2011 Jun 28. PMID 21712482
- [Background] Kim JS, Zee DS. Clinical practice. Benign paroxysmal positional vertigo. N Engl J Med. 2014 Mar 20;370(12):1138-47. doi: 10.1056/NEJMcp1309481. No abstract available. PMID 24645946
- [Background] Hoffer ME, Gottshall KR, Moore R, Balough BJ, Wester D. Characterizing and treating dizziness after mild head trauma. Otol Neurotol. 2004 Mar;25(2):135-8. doi: 10.1097/00129492-200403000-00009. PMID 15021772
- [Background] Hilton M, Pinder D. The Epley manoeuvre for benign paroxysmal positional vertigo--a systematic review. Clin Otolaryngol Allied Sci. 2002 Dec;27(6):440-5. doi: 10.1046/j.1365-2273.2002.00613.x. PMID 12472509
- [Background] Brodsky, J.R., Cusick, B.A., Zhou, G. Delayed diagnosis and treatment of benign paroxysmal positioning vertigo (BPPV) in children and adolescents with post-concussive syndrome. Poster presentation at the Triological Society Meeting, Miami, FL, 2016.